CLINICAL TRIAL: NCT05467319
Title: Feasibility and Efficacy of Intravenous Ferric Derisomaltose to Correct Pre-operative Iron-deficiency Anemia in Patients Undergoing Gynecologic Oncology Surgery: a Pilot Randomized Double Blinded Parallel Group Placebo-controlled Study
Brief Title: Ferric Derisomaltose/Iron Isomaltoside and Outcomes in the Recovery of Gynecologic Oncology ERAS
Acronym: FORGE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alberta Health Services, Calgary (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Principal Investigator, Steven Bisch, Principal Investigator, Alberta Health Services, Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FORGEII
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Gynecologic Cancer; Anemia, Iron Deficiency; Surgery
Keywords: Ferric derisomaltose; iron isomaltoside; intravenous iron
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric derisomaltose; iron isomaltoside 1000; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel groups, randomized placebo-controlled, double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Intravenous treatment will be prepared by an unblinded provider and placed in opaque bags/tubing to blind the patient, administrator of the medication, and subsequent outcome assessors and care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric derisomaltose (Experimental): 1000mg of intravenous Ferric derisomaltose/Iron isomaltoside in 100mL of normal saline will be administered 21-90 days prior to planned surgery for gynecologic malignancy as a single dose.
  Interventions: Drug: Ferric Derisomaltose Injection
- Placebo (Placebo Comparator): 100mL of normal saline will be administered 21-90 days prior to planned surgery for gynecologic malignancy as a single dose.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ferric Derisomaltose Injection — 1000mg of ferric derisomaltose in 100mL of normal saline by intravenous infusion
  Other Names: iron isomaltoside; Monoferric; Monofer
  Arms: Ferric derisomaltose
Drug: Normal saline — 100 mL of 0.9% normal saline (w/v) by intravenous infusion
  Arms: Placebo

SUMMARY:
Iron deficiency has been reported in up to 35% of patients with a gynecologic malignancy. These patients often require surgical intervention to determine the stage and to treat their illness. Blood transfusions occur in approximately 14% of these surgeries and carry immediate and long-term risks, including surgical site infection, cancer recurrence, and increased surgical length of stay. Intravenous iron formulations have the potential to rapidly correct anemia in patients with gynecologic malignancy and potentially decrease blood transfusion and complications following surgery. This prospective, randomized, placebo-controlled, double blind study aims to assess the effectiveness of preoperative ferric derisomaltose/iron isomaltoside compared to placebo in correcting preoperative hemoglobin in patients undergoing surgery for gynecologic malignancy. The primary outcome is to assess the effectiveness of this formulation on pre-operative hemoglobin, and the feasibility of a larger, outcomes based, study in the future. Exploratory outcomes are to assess the effect of preoperative intravenous iron on surgical length of stay, complications, and patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and signed written informed consent
2. Patients undergoing elective major surgery on the gynecologic oncology service with the following criteria will be considered for inclusion:

   1. The indication for the operation may be for suspected or proven gynecologic malignancy.
   2. Major surgery is defined as an operation of a duration of 1 hour or greater, with an Aletti complexity score of at least 1[19].
   3. The expected time from recruitment to surgery is at least 28 days.
3. Screening haemoglobin less than 120g/L and transferrin saturation (TSAT) <20%
4. Randomization and administration of study infusion a minimum of 21 days and maximum 90 days before planned operation.
5. Negative pregnancy test for women of childbearing potential (within last 7 days), and agree to use effective form of contraception until 6 weeks post treatment (if applicable)
6. Laboratory data used for determination of eligibility at the baseline visit must not be older than 4 weeks.

Exclusion Criteria:

1. Known history of acquired iron overload, or family history of haemochromatosis or thalassemia, or TSAT >50%
2. Known alternative cause for anemia (e.g. B12 or folate deficiency, or haemoglobinopathy)
3. Known hypersensitivity to FDI or its excipients
4. Temperature >38 C or patient on non-prophylactic antibiotics
5. Known chronic liver disease or active hepatitis
6. Received erythropoietin or IV iron therapy in previous 12 weeks
7. If LFT's are ordered, either clinically indicated or for chemotherapy, and screening alanine transaminase (ALT) or aspartate transaminase (AST) is above three times the upper limit of normal (ULN) range
8. Immunosuppressive therapy (for solid organ transplant), or renal dialysis (current, or planned within next 12 months)
9. Unfit for elective surgery
10. Pregnancy or lactation
11. Unable to fully comprehend and/or perform study procedures
12. Cervical cancer with a clinical stage of 2A or greater.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative hemoglobin level | 0 to 3 days prior to planned surgical intervention
  Hemoglobin measured, in g/L, following intervention prior to planned gynecologic surgery.

IPD SHARING:
Plan to Share IPD: Undecided